CLINICAL TRIAL: NCT02442791
Title: GLP-1 Analogs for Neuroprotection After Out-of-hospital Cardiac Arrest, a Randomized Clinical Trail
Brief Title: GLP-1 Analogs for Neuroprotection After Cardiac Arrest
Acronym: GLIP1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jesper Kjaergaard (Other)
Responsible Party: Sponsor-Investigator, Jesper Kjaergaard, MD, DMSc, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-TTMPharma-001
Record Dates: First submitted 2015-01-25; First posted 2015-05-13 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Cardiac Arrest; Coma
Keywords: Cardiac arrest; GLP-1; Neuroprotection
MeSH Terms: conditions — Heart Arrest; Coma | interventions — Exenatide; Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GLP-1 (Experimental): Half of the participants will receive the study drug, that will be given as follows:
  250 mL isotonic sodium chloride added 1.5 mL of 20% Human Albumin added 25 microg Byetta (Lilly, Exenatide).
  The study drug infusion is initiated as soon as possible at rate of 72ml/hour (0.12 μg/min) for 15 min (set volume at 18 ml), followed by 26ml/hour (0.043 μg/min) to be continued for 6 hours (set volume at 156 ml). This concludes the pharmacological intervention.
  Interventions: Drug: Byetta (Lilly, Exenatide); Other: 20% Human Albumin
- Placebo (Placebo Comparator): Half of the participants will receive placebo, that will be given as follows:
  250 mL isotonic sodium chloride added 1.5 mL of 20% Human Albumin. The placebo infusion is administered exactly the same way as the study drug infusion.
  Interventions: Other: 20% Human Albumin

INTERVENTIONS:
Drug: Byetta (Lilly, Exenatide) — See description of Arms
  Other Names: Byetta
  Arms: GLP-1
Other: 20% Human Albumin — See description of Arms

SUMMARY:
Experimental studies and previous clinical trials suggest neuroprotective effects of GLP-1 analogs in various degenerative neurological diseases, and in hypoxic brain injuries in experimental designs. This study is designed as a safety and feasibility study with patients randomized 1:1 to receive GLP-1 analogs immediately after hospital admission after out of hospital cardiac arrest.

DETAILED DESCRIPTION:
In comatose patients resuscitated from out of hospital cardiac arrest, neurological injuries remain the leading cause of death. The in-hospital mortality is reported at 30-50%, and the total mortality, although improved substantially over the last decade, remain to be significant, in most countries up to 90%. The brain of a patient resuscitated after cardiac arrest (CA) may have suffered ischemia and when the spontaneous circulation is re-established, the subsequent reperfusion may cause further damage. Brain ischemia and the reperfusion injury lead to tissue degeneration and loss of neurological function, the extent dependent on duration and density of the insult. Temperature control and mild induced hypothermia (MIH) (33-36°C) mitigate this damage in the experimental setting and clinical trials have shown promising results in improving neurological function and survival. Recent large scale clinical trials however have investigated milder degree of hypothermia in this setting, which suggest a role for active neuroprotection outside of temperature management. Also recently, increased attention to the possible role of Glucagon-Like Peptide-1 (GLP-1) in neuroprotection has been raised, both in the context of ameliorating degenerative disease and in reducing inflammation on ischemic cerebral stroke.

Several experimental studies have shown that GLP-1 analogs has a beneficial effect in the treatment of various degenerative neurological diseases such as Alzheimer's disease and Parkinson's disease. GLP-1 analogs have been shown to reduce brain infarct size in mice after focal brain ischemia as well as to reduce heart infarct size in swine in a model of myocardial infarction.

Recent clinical testing in humans have demonstrated a benefit of GLP-1 infusion on myocardial infarct size and a larger salvage index in patients with myocardial infarction. The GLP-1 analogs were infused in acutely ill patients in many ways similar to cardiac arrest patients with no increased risk of adverse events.

This study is a double blinded randomized study seeking to evaluate the potential neuroprotective effects of GLP-1 analogs infused in comatose patients after out of hospital cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* Out of hospital cardiac arrest (OHCA) of presumed cardiac cause
* Sustained return of spontaneous circulation (ROSC)
* Unconsciousness (GCS <8 (Glasgow coma scale)) (patients not able to obey verbal commands)
* Sustained ROSC (Sustained ROSC: Sustained ROSC is when chest compressions have been not required for 20 consecutive minutes and signs of circulation persist)

Exclusion Criteria:

* Conscious patients (obeying verbal commands)
* Females of childbearing potential (unless a negative pregnancy test can rule out pregnancy within the inclusion window)
* In-hospital cardiac arrest (IHCA)
* OHCA of presumed non-cardiac cause, e.g. after trauma or dissection/rupture of major artery OR Cardiac arrest caused by initial hypoxia (i.e. drowning, suffocation, hanging).
* Known bleeding diathesis (medically induced coagulopathy (e.g. warfarin, clopidogrel) does not exclude the patient).
* Suspected or confirmed acute intracranial bleeding
* Suspected or confirmed acute stroke
* Unwitnessed asystole
* Known limitations in therapy and Do Not Resuscitate-order
* Known disease making 180 days survival unlikely
* Known pre-arrest cerebral performance category 3 or 4
* >4 hours (240 minutes) from ROSC to screening
* Systolic blood pressure <80 mm Hg in spite of fluid loading/vasopressor and/or inotropic medication/intra aortic balloon pump/axial flow device*
* Temperature on admission <30°C.
* Known allergy to GLP-1 analogs, including Exenatide
* Known pancreatitis
* Diabetic ketoacidosis,
* Uncorrected blood glucose at admission < 2.5 mmol/l.

  * If the systolic blood pressure (SBP) is recovering during the inclusion window (220 minutes) the patient can be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Feasibility: Over 90% initiation of study drug infusion | 4 hours from return of spontaneous circulation
Efficacy assessed by Area under the Neuron-specific Enolase curve | 72 hours from admission

SECONDARY OUTCOMES:
Neurological prognostication | Day 5
  Blinded neurological evaluation by neurologist on "VAS-scale"
Area under Neuron-specific Enolase curves (NSE) | 48 hours
  Daily measurements of NSE values
All cause mortality | 180 days
  Vital status by end of study by registry based follow-up
Cerebral status | 30 days, 90 days and 180 days
  Telephone based assessment of Cerebral Performance Category and modified Rankin Scale.
Safety: Cumulated incidence of serious adverse events related to study drug: death, need for mechanical hemodynamic support, hypoglycaemia < 3.0 mmol/l, pancreatitis (S-amylase > 3 UNL), need for renal replacement therapy in the first 3 days. | 180 days
Area under S100b curve | 48 hours
  Daily measurements of S100b

OTHER OUTCOMES:
Left Ventricular Ejection Fraction (LVEF) | Day 5 or later
  LVEF on last in-hospital echocardiogram.
EEG findings | Day 3 to 5
  Presence of EEG findings associated with poor prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Kjaergaard, MD., DMSc., Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Kardiologisk Afdeling, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Result] Wiberg S, Hassager C, Schmidt H, Thomsen JH, Frydland M, Lindholm MG, Hofsten DE, Engstrom T, Kober L, Moller JE, Kjaergaard J. Neuroprotective Effects of the Glucagon-Like Peptide-1 Analog Exenatide After Out-of-Hospital Cardiac Arrest: A Randomized Controlled Trial. Circulation. 2016 Dec 20;134(25):2115-2124. doi: 10.1161/CIRCULATIONAHA.116.024088. Epub 2016 Nov 12. PMID 27838646
- [Derived] Toftgaard Pedersen A, Kjaergaard J, Hassager C, Frydland M, Hartvig Thomsen J, Klein A, Schmidt H, Moller JE, Wiberg S. Association between inflammatory markers and survival in comatose, resuscitated out-of-hospital cardiac arrest patients. Scand Cardiovasc J. 2022 Dec;56(1):85-90. doi: 10.1080/14017431.2022.2074093. PMID 35546563
- [Derived] Wiberg S, Kjaergaard J, Schmidt H, Thomsen JH, Frydland M, Winther-Jensen M, Lindholm MG, Hofsten DE, Engstrom T, Kober L, Moller JE, Hassager C. The Glucagon-Like Peptide-1 Analog Exenatide Increases Blood Glucose Clearance, Lactate Clearance, and Heart Rate in Comatose Patients After Out-of-Hospital Cardiac Arrest. Crit Care Med. 2018 Feb;46(2):e118-e125. doi: 10.1097/CCM.0000000000002814. PMID 29189347
- [Derived] Wiberg S, Hassager C, Thomsen JH, Frydland M, Hofsten DE, Engstrom T, Kober L, Schmidt H, Moller JE, Kjaergaard J. GLP-1 analogues for neuroprotection after out-of-hospital cardiac arrest: study protocol for a randomized controlled trial. Trials. 2016 Jun 30;17(1):304. doi: 10.1186/s13063-016-1421-2. PMID 27363489